CLINICAL TRIAL: NCT05562648
Title: Comparison of the Efficacy of Manual Therapy Techniques and Electrotherapy Modalities in Individuals With Non-specific Low Back Pain
Brief Title: Efficacy of Manual Therapy Techniques and Electrotherapy Modalities in Individuals With Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: back pain
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Back Pain
Keywords: manuel therapy
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy techniques (Experimental): Myofascial release is a soft tissue method that provides removal of adhesions and tissue tension in tissues due to overload and repetitive use. These adhesions and unbalanced tissue tensions in the tissues can cause muscle weakness, numbness, pain, tingling and burning sensation. The soft tissue is palpated by the physiotherapist and pressure is applied directly to the skin until the tissue barrier is felt in the direction of restriction. Once the tissue barrier is present, it is applied for 90-120 seconds, without slipping on the skin or forcing the tissue, until the fascia complex begins to loosen and a softening sensation is achieved.
  Interventions: Other: Manual therapy techniques
- Electrophysical agents (Active Comparator): Evidence levels for approaches commonly used in the clinic for the treatment of chronic low back pain were generally very low to moderate. TENS (Transcutaneous Electrical Nerve Stimulation) is the most preferred application in the treatment of chronic pain in patients who receive conventional treatment in the clinic. TENS is a physiotherapy modality used to inhibit pain by stimulating the sensory nerves by applying a low frequency electrical current.
  Interventions: Other: Electrophysical agents

INTERVENTIONS:
Other: Manual therapy techniques — Myofascial trigger points are determined and the physiotherapist applies a light and continuous local pressure on them with his/her finger, usually not more than 30 seconds, until the moment of muscle relaxation, and as a result, the pain is expected to decrease to 0 (zero) and he withdraws his finger. He can do 3-5 repetitions until he sees relaxation in the muscle and reduction/disappearance of the pain.
  Spinal mobilization is defined as low-speed, non-trust, passive movement within or at the limit of joint range of motion. Mobilization is low-speed, non-trust, passive joint movement.
  MUSCLE ENERGY TECHNIQUES The muscle energy technique is a treatment technique that includes alternating periods of resistant muscle contractions and active-assist stretching, mostly used by osteopaths, physiotherapists, and chiropractors.
  Arms: Manual therapy techniques
Other: Electrophysical agents — TENS TENS is a low-frequency electrical current applied to the stimulation of sensory nerves, used for the inhibition of pain sensation. Pain inhibition of TENS is based on 3 basic mechanisms. These; gate control mechanism (segmental inhibition), release of endogenous opioids and reduction of excitability with repetitive stimulation (inhibition from pattern).
  Ultrasound is an effective electrotherapy modality with a deep heating feature. In addition, it has been suggested that the analgesic effect of ultrasound occurs with the stimulation of sensory afferents and the activation of the gate control mechanism in the posterior horn of the spinal cord.
  Arms: Electrophysical agents

SUMMARY:
Low back pain is the fifth most common reason for doctor visits, affecting about 60-80% of people in their lifetime. Despite this, there are not enough diagnostic and treatment methods in the literature to fully elucidate non-specific low back pain. In this case, the research showed that non-specific low back pain should be handled with a biopsychosocial approach, and its relationship with fascia and myofascial meridians should be investigated.

DETAILED DESCRIPTION:
According holistic that approach patients with non-specific low back pain. Instead of examining the problem of low back pain in the society only in the form of muscles, joints, ligaments, etc.; should evaluate low back pain over the fascia. It is seen that most studies in the literature only examine the painful area and tissue problems in its immediate vicinity, and therefore they approach low back pain with symptomatic treatment. In recent studies, however, the main problem is not limited to the painful area only; It has been determined that the tissue response caused by the problems in different parts of the body is transmitted to more distant regions via the fascia and myofascial meridians.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-60
* Volunteering to work
* The person has a complaint of low back pain for more than 3 months
* Diagnosis of chronic low back pain by the doctor
* Being able to read and write and be cooperative.
* Not having received treatment for the lumbar region in the last 3 months
* having an MRI in the last 6 months.

Exclusion Criteria:

* Not having any lumbar surgery or vertebral fracture
* Having neurological, radiculopathy, inflammatory, etc. disease
* Having spinal deformities such as scoliosis, kyphosis
* Having a vestibular or respiratory disorder
* Having auditory or cognitive impairment
* Medication that will affect the balance (sedatives, etc.)
* Patients with lower extremity amputation
* Those who want to quit working during the study period, those who do not attend regularly.
* Conditions such as cancer, infection, etc. in the spinal region

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 4 weeks
  It is a questionnaire to evaluate the disability levels and quality of life faced by patients due to low back pain. It was developed to evaluate pain-related limitation in people with acute, subacute, or chronic low back pain. It includes 1 item related to pain and 9 items related to activities of daily living (personal care, lifting, walking, sitting, sanding, sleep, sexual life, social life and travel). Each item is measured on a 6-point rank scale between 0 and 5 points according to the scenarios it contains. At the end of the survey, the scores are summed and the percentage value is calculated for the total score.
Beck Depression Scale | 4 weeks
  This scale has been shown to accurately measure the level of depression. The scale consists of 21 questions with 4 options, each corresponding to 0-3 points, and the patient is asked to choose the appropriate sentence according to his condition in the last week. mood, pessimism, sense of failure, dissatisfaction, sense of guilt, sense of punishment, self-hatred, self-blame, desire for self-punishment, crying spells, irritability, social introversion, indecisiveness, deterioration of body perception, determination of workability, sleep disorders, 21 symptoms and behaviors including fatigue, fatigue, decreased appetite, weight loss, somatic complaints and loss of libido are questioned.
Pittsburgh Sleep Survey Index: | 4 weeks
  The Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality and disturbance over the past 1-month time period. This questionnaire has seven scales including Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency (the ratio of sleep time to time in bed), Sleep Disorders (waking up at night), Sleeping Medication Use, and Daytime Dysfunction (problems caused by insomnia during the day). . Calculation of scores for these seven components yields a final score. The score for each scale ranges from 0-3, with three points on each scale indicating the maximum negative value. The total score of this questionnaire is between 0-21, and a total score greater than 5 is an indication of inadequate sleep quality.
Modified Schober Test: | 4 weeks
  It is another method used to evaluate the flexibility/mobility of the lumbar spine. While the patient is standing in an upright position, the lumbosacral junction determined in accordance with the two sacroiliac joint positions is marked with a pencil. The second point is marked 5 cm below this marked point, and the third point is marked 10 cm above it. Afterwards, the patient is asked to flex the trunk as much as possible while the knees are in full extension. After the movement is completed, the newly formed distance between the second and third points is measured in "cm" with the help of a tape measure. Subtract 15 cm from the value obtained from the measurement result, and if the calculation is less than 7 cm, it is assumed that the lumbar flexibility has decreased.

SECONDARY OUTCOMES:
The Visual Analog Scale (VAS) | 4 weeks
  The Visual Analog Scale (VAS) was used to evaluate the pain intensity of patients with low back pain during movement and rest. According to the VAS, patients are asked to indicate their pain intensity by giving a number from 1 to 10, with a score of "0" if the pain sensation is no pain, and "10" if the pain sensation is the most severe.
Fingertip-to-Floor Test | 4 weeks
  While the patient is standing in an upright position, the patient is asked to flex the trunk as much as possible without flexing the knees, with the hands free. The distance between the third finger of the patient and the ground is recorded with the help of a tape measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol hospital, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: data — https://pubmed.ncbi.nlm.nih.gov/21943614/ — Rozzi, P., Bongiorno, D., & Vitturini, C. (2011). Fascial release effects on patients with non-specific cervical or lumbar pain. Journal of bodywork and movement therapies, 15(4), 405-416.